CLINICAL TRIAL: NCT03906669
Title: A Window of Opportunity Study of Endocrine Therapy With and Without Prometrium in Postmenopausal Women With Early Stage Hormone Receptor-positive Breast Cancer.
Brief Title: A Window of Opportunity Study of Pre-operative Endocrine Therapy With and Without Prometrium in Postmenopausal Women With Early Stage Breast Hormone Receptor Positive (HR+) Human Epidermal Receptor 2 Negative (HER2-) Breast Cancer.
Acronym: WinPro
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St Vincent's Hospital (Other)
Responsible Party: Principal Investigator, Elgene Lim, Associate Professor, St Vincent's Hospital, Sydney
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTRN1261000928213
Record Dates: First submitted 2018-09-18; First posted 2019-04-08 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Early-stage Breast Cancer; Hormone Receptor Positive Tumor
Keywords: early stage breast cancer; prometrium; progesterone; post-menopausal; endocrine therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; Progesterone; Tamoxifen

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Letrozole (Active Comparator): Letrozole 2.5mg PO daily for 14 days between diagnosis of breast cancer and definite surgery
  Interventions: Drug: Letrozole
- Letrozole and Prometrium (Experimental): Letrozole 2.5mg PO daily and Prometrium 300mg PO daily for 14 days between diagnosis of breast cancer and definite surgery
  Interventions: Drug: Letrozole and Prometrium
- Tamoxifen and Prometrium (Experimental): Tamoxifen 20mg PO daily and Prometrium 300mg PO daily for 14 days between diagnosis of breast cancer and definite surgery
  Interventions: Drug: Tamoxifen and Prometrium

INTERVENTIONS:
Drug: Letrozole — PO daily for 14 days
  Arms: Letrozole
Drug: Letrozole and Prometrium — PO daily for 14 days
  Arms: Letrozole and Prometrium
Drug: Tamoxifen and Prometrium — PO daily for 14 days
  Arms: Tamoxifen and Prometrium

SUMMARY:
A phase II randomised, open label study of pre-operative endocrine therapy with & without prometrium in postmenopausal women with early stage breast hormone receptor positive (HR+) human epidermal receptor 2 negative (HER2-) breast cancer.

DETAILED DESCRIPTION:
There is bidirectional interplay between the progesterone receptor (PR) and oestrogen receptor (ER) in human breast cancers. There is evidence for a reprogramming of ER chromatin binding sites with 470 genes differentially regulated by dual treatment with estrogen plus progestogen compared to estrogen alone in breast cancer cell lines. Functionally, there was an additive anti-cancer effect with the addition of natural progesterone to endocrine therapy in preclinical breast cancer models.

This is a phase II multi-site, randomised, open-label, three-arm, study in 200 postmenopausal women with early-stage ER+, PR+, HER2-negative breast cancer. Eligible patients will be randomised (1:1:1) to receive 14 days of intervention with either letrozole 2.5mg PO daily (arm 1), letrozole 2.5mg + prometrium 300mg PO daily (arm 2) or tamoxifen 20mg + prometrium 300mg PO daily (arm 3), between diagnosis of breast cancer and definitive surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed ER+ and PR+ breast cancer (defined as ≥10% positive staining cells)
2. Histologically confirmed HER2-negative breast cancer (defined as IHC 0-1 and/or FISH/CISH <2.2)
3. Tumour size ≥1 cm as measured by ultrasound and/or mammogram
4. Ability to understand all patient information and informed-consent documents, written informed consent to participate in the trial, and to avail tissue and blood samples for research
5. Aged 18 years or older

Exclusion Criteria:

1. Women currently on hormone therapies, including hormone replacement therapy and oral contraceptive pill
2. Locally advanced/inoperable and inflammatory breast cancer
3. Planned for a mastectomy (due to increased risk of venous thromboembolism)
4. Clinical evidence of metastatic disease
5. Patients treated with other preoperative systemic therapies
6. Nut allergy (prometrium contains peanut oil)
7. Prior history of uterine cancer, deep vein thrombosis, pulmonary embolism or clotting disorder
8. Women who are pregnant or breast-feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-03-20 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Geometric mean suppression of proliferation marker Ki67 | After two weeks of intervention, compared with baseline
  The geometric mean suppression of the centrally assessed proliferation marker Ki67, after two weeks of intervention, compared with baseline

SECONDARY OUTCOMES:
Safety and tolerability: number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 2 years
  Safety and tolerability of combination therapy (NCI-CTCAE v4.0)

OTHER OUTCOMES:
Define a gene set as a predictive biomarker for a reduction in Ki67 | 4 years
  Expression of gene signature will be tested in the pre- and post-intervention tissues using the Nanostring nCounter system
Evaluate changes in the apoptotic markers Bcl-2 and Caspase 3 in the tumors following intervention | 4 years
  Immunohistochemistry of the pre and post intervention tissue samples
Evaluate changes in ER, PR, AR, FoxA1, Cyclin D1 protein and mRNA expression in the tumors following intervention | 4 years
  Immunohistochemistry of the pre and post intervention tissue samples

CONTACTS AND LOCATIONS:
Overall Officials: Elgene Lim, MBBS FRACP PhD, Principal Investigator — Garvan Research Institute
Locations (1):
- St Vincent's Hospital, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mohammed H, Russell IA, Stark R, Rueda OM, Hickey TE, Tarulli GA, Serandour AA, Birrell SN, Bruna A, Saadi A, Menon S, Hadfield J, Pugh M, Raj GV, Brown GD, D'Santos C, Robinson JL, Silva G, Launchbury R, Perou CM, Stingl J, Caldas C, Tilley WD, Carroll JS. Progesterone receptor modulates ERalpha action in breast cancer. Nature. 2015 Jul 16;523(7560):313-7. doi: 10.1038/nature14583. Epub 2015 Jul 8. PMID 26153859
- [Background] Lim E, Tarulli G, Portman N, Hickey TE, Tilley WD, Palmieri C. Pushing estrogen receptor around in breast cancer. Endocr Relat Cancer. 2016 Dec;23(12):T227-T241. doi: 10.1530/ERC-16-0427. Epub 2016 Oct 11. PMID 27729416